CLINICAL TRIAL: NCT03088072
Title: A Pilot Study of Edoxaban in Patients With Non-Valvular Atrial Fibrillation and Left Atrial Appendage Closure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Health (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Matthew J Price, Principal Investigator, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17-6931
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Non-Valvular Atrial Fibrillation; Left Atrial Appendage Closure
Keywords: Edoxaban; WATCHMAN device
MeSH Terms: interventions — edoxaban; Aspirin; Clopidogrel; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Edoxaban Arm (Other): All patients enrolled in the study will receive 6 weeks of edoxaban therapy, at which time a TEE will be performed. If the result is acceptable, edoxaban will be discontinued, and the patient will be treated with dual antiplatelet therapy (aspirin and clopidogrel) until 6 month follow-up. If device thrombus is present at 6 week TEE, patient will be transitioned to aspirin and adjusted-dose warfarin and LAA reassessed by TEE in 6 weeks; further warfarin will be continued according to operator preference. Subjects will have a 6 month follow-up visit prior to study completion. After study completion, patients may be treated with aspirin monotherapy according to the FDA instructions for use for the WATCHMAN device, or according to operator discretion.
  Interventions: Drug: Edoxaban; Device: WATCHMAN LAA Closure; Drug: Aspirin and Clopidogrel; Drug: Aspirin and Warfarin

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 60mg once daily in patients with CrCl >50- ≤95 mL/min, or 30mg once daily in patients with CrCL 15-50 mL/min.
  If at 6 week TEE LAA closure is deemed acceptable by the operator (i.e., peri-device flow <5mm), edoxaban will be discontinued. Aspirin 81mg daily and clopidogrel 75mg daily will be administered until 6-month follow-up, then clopidogrel will be discontinued.
  If LAA unacceptable on 6-week TEE due to peri-device flow ≥5mm, edoxaban will be continued for an additional 6 weeks, and LAA reassessed by TEE If device thrombus is present at 6-week TEE, patient will be transitioned to aspirin 81 mg daily and adjusted-dose warfarin (goal INR, 2.0-3.0), and LAA reassessed by TEE in 6 weeks; further warfarin will be continued according to operator preference.
  Other Names: Savaysa
Device: WATCHMAN LAA Closure — Per Inclusion Criteria, enrolled subjects must have a successful Left Atrial Appendage (LAA) Closure using the WATCHMAN Device
Drug: Aspirin and Clopidogrel — If at 6 week TEE LAA closure is deemed acceptable by the operator edoxaban will be discontinued, and aspirin 81mg daily and clopidogrel 75mg daily will be administered until 6-month follow-up. Then clopidogrel will be discontinued.
  Aspirin 325mg daily rather than 81mg daily can be administered according to operator preference after the 6-week follow-up visit.
Drug: Aspirin and Warfarin — If device thrombus is present at 6-week TEE, patient will be transitioned to aspirin 81 mg daily and adjusted-dose warfarin (goal INR, 2.0-3.0), and LAA reassessed by TEE in 6 weeks; further warfarin will be continued according to operator preference.

SUMMARY:
This is a single arm, open label, single site study assessing the feasibility of post-procedural edoxaban therapy in atrial fibrillation (AF) patients after clinically indicated WATCHMAN left atrial appendage (LAA) closure.

DETAILED DESCRIPTION:
This is a single site, PI initiated pilot study. This study will enroll up to 75 patients who are clinically indicated for a Left Atrial Appendage (LAA) closure with the commercially available WATCHMAN device. Subjects will be enrolled if they meet study inclusion/exclusion criteria and have a successful LAA closure. All patients enrolled in the study will receive 6 weeks of edoxaban therapy. At 6 weeks post LAA closure a Transesophageal Echocardiography (TEE) will be performed. If the result is acceptable, edoxaban will be discontinued and the patient will be treated with dual antiplatelet therapy (aspirin and clopidogrel) until 6 month follow-up. After study completion, patients may be treated with aspirin monotherapy according to the FDA instructions for use for the WATCHMAN device, or according to operator discretion.

ELIGIBILITY:
Inclusion Criteria:

* The patient has documented paroxysmal, persistent, or permanent non-valvular AF (i.e., the patient has not been diagnosed with rheumatic mitral valve disease).
* LAA closure with the WATCHMAN device is planned
* The patient fulfills the FDA indication for WATCHMAN LAA closure
* The patient or legal representative is able to understand and willing to provide written informed consent to participate in the trial
* The patient is able and willing to return for required follow-up visits and examinations.
* The patient is 18 years of age or older

Exclusion Criteria:

* Conditions other than atrial fibrillation that require anti-coagulation (e.g., a prosthetic heart valve)
* Stroke within the previous 7 days
* Hypersensitivity to edoxaban
* Moderate or severe mitral stenosis
* A need for aspirin at a dose of >81 mg a day
* A need for on-going treatment with dual antiplatelet therapy with aspirin and clopidogrel
* A need for on-going treatment with ticagrelor or prasugrel
* No LAA closure device implanted during procedure
* Procedural complication of LAA closure (e.g., stroke, systemic embolism, bleeding, vascular complication [e.g., groin hematoma >10cm, AV fistula, or pseudoaneurysm), or serious pericardial effusion)
* Planned surgery or invasive procedure within 6±2 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Death, stroke, systemic embolism or GUSTO outcomes | 6 weeks
  Composite of death, stroke, systemic embolism, or GUSTO moderate/severe bleeding will be collected at 6 weeks post-WATCHMAN LAA closure

SECONDARY OUTCOMES:
Death, stroke, or systematic embolism outcomes | 6 weeks and 6 months
  Composite of death, stroke, or systemic embolism at 6 weeks and 6 months
Death, stroke, or systematic embolism or GUSTO outcomes | 6 months
  Composite of death, stroke, systemic embolism or GUSTO moderate/severe bleeding at 6 months
Device thrombus oucomes | 6 weeks
  TEE-confirmed device thrombus (according to core laboratory) at 6 weeks
TEE peri-device flow outcomes | 6 weeks
  Rate of peri-device flow >=5mm at 6 week follow-up TEE
GUSTO mild, moderate, severe, and GUSTO moderate/severe bleeding outcomes | 6 weeks and 6 months
  Individual endpoints of GUSTO mild, moderate, severe, and GUSTO moderate/severe bleeding at 6 weeks and 6 months
Premature discontinuation rate of study drug | 6 weeks
  Premature discontinuation rate of study drug before 6-week visit
Bleeding outcomes | 6 weeks and 6 months
  Bleeding according to the months Bleeding Academic Research Consortium (BARC) criteria at 6 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Price, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Price MJ, Valderrabano M. Left atrial appendage closure to prevent stroke in patients with atrial fibrillation. Circulation. 2014 Jul 8;130(2):202-12. doi: 10.1161/CIRCULATIONAHA.114.009060. No abstract available. PMID 25001625
- [Background] Price MJ, Holmes DR. Mechanical closure devices for atrial fibrillation. Trends Cardiovasc Med. 2014 Aug;24(6):225-31. doi: 10.1016/j.tcm.2014.06.001. Epub 2014 Jun 8. PMID 25066488
- [Background] Xu H, Ruff CT, Giugliano RP, Murphy SA, Nordio F, Patel I, Shi M, Mercuri M, Antman EM, Braunwald E. Concomitant Use of Single Antiplatelet Therapy With Edoxaban or Warfarin in Patients With Atrial Fibrillation: Analysis From the ENGAGE AF-TIMI48 Trial. J Am Heart Assoc. 2016 Feb 23;5(2):e002587. doi: 10.1161/JAHA.115.002587. PMID 26908401
- [Background] Dans AL, Connolly SJ, Wallentin L, Yang S, Nakamya J, Brueckmann M, Ezekowitz M, Oldgren J, Eikelboom JW, Reilly PA, Yusuf S. Concomitant use of antiplatelet therapy with dabigatran or warfarin in the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) trial. Circulation. 2013 Feb 5;127(5):634-40. doi: 10.1161/CIRCULATIONAHA.112.115386. Epub 2012 Dec 27. PMID 23271794
- [Background] Lamberts M, Gislason GH, Lip GY, Lassen JF, Olesen JB, Mikkelsen AP, Sorensen R, Kober L, Torp-Pedersen C, Hansen ML. Antiplatelet therapy for stable coronary artery disease in atrial fibrillation patients taking an oral anticoagulant: a nationwide cohort study. Circulation. 2014 Apr 15;129(15):1577-85. doi: 10.1161/CIRCULATIONAHA.113.004834. Epub 2014 Jan 27. PMID 24470482
- [Background] Price MJ, Reddy VY, Valderrabano M, Halperin JL, Gibson DN, Gordon N, Huber KC, Holmes DR Jr. Bleeding Outcomes After Left Atrial Appendage Closure Compared With Long-Term Warfarin: A Pooled, Patient-Level Analysis of the WATCHMAN Randomized Trial Experience. JACC Cardiovasc Interv. 2015 Dec 28;8(15):1925-1932. doi: 10.1016/j.jcin.2015.08.035. Epub 2015 Nov 25. PMID 26627989
- [Background] Lopes RD, Al-Khatib SM, Wallentin L, Yang H, Ansell J, Bahit MC, De Caterina R, Dorian P, Easton JD, Erol C, Ezekowitz JA, Gersh BJ, Granger CB, Hohnloser SH, Horowitz J, Hylek EM, McMurray JJ, Mohan P, Vinereanu D, Alexander JH. Efficacy and safety of apixaban compared with warfarin according to patient risk of stroke and of bleeding in atrial fibrillation: a secondary analysis of a randomised controlled trial. Lancet. 2012 Nov 17;380(9855):1749-58. doi: 10.1016/S0140-6736(12)60986-6. Epub 2012 Oct 2. PMID 23036896
- [Background] Bosche LI, Afshari F, Schone D, Ewers A, Mugge A, Gotzmann M. Initial Experience With Novel Oral Anticoagulants During the First 45 Days After Left Atrial Appendage Closure With the Watchman Device. Clin Cardiol. 2015 Dec;38(12):720-4. doi: 10.1002/clc.22478. Epub 2015 Oct 14. PMID 26467851
- [Background] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Background] ACTIVE Writing Group of the ACTIVE Investigators; Connolly S, Pogue J, Hart R, Pfeffer M, Hohnloser S, Chrolavicius S, Pfeffer M, Hohnloser S, Yusuf S. Clopidogrel plus aspirin versus oral anticoagulation for atrial fibrillation in the Atrial fibrillation Clopidogrel Trial with Irbesartan for prevention of Vascular Events (ACTIVE W): a randomised controlled trial. Lancet. 2006 Jun 10;367(9526):1903-12. doi: 10.1016/S0140-6736(06)68845-4. PMID 16765759
- [Background] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Price MJ. Left atrial appendage occlusion with the WATCHMAN for stroke prevention in atrial fibrillation. Rev Cardiovasc Med. 2014;15(2):142-51. doi: 10.3909/ricm0733. PMID 25051131